CLINICAL TRIAL: NCT02087332
Title: Randomized Open-label Comparative Study of Britomar (Prolonged Release Torasemide) and Diuver (Torasemide) to Assess Effects on Natriuresis and Central Hemodynamics in Patients With Arterial Hypertension and Chronic Heart Failure
Brief Title: Investigator Initiated Randomized Open-label Comparative Study of Britomar (Prolonged Release Torasemide) and Diuver (Torasemide) to Assess Effects on Natriuresis and Central Hemodynamics.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Society of Specialists in Heart Failure (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOR-IIT-001; TOR-IIT-001 (Other Grant/Funding Number: Investigator Initiated study. Grant was provided by Takeda Pharmaceuticals LLC, Russia)
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Arterial Hypertension; Chronic Heart Failure
Keywords: Kidney damage hypertension cardiovascular diseases, congestive heart failure renal function natriuresis natriuresis monitoring
MeSH Terms: conditions — Hypertension | interventions — Torsemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prolonged release Torasemide (Britomar) (Experimental): Prolonged release Torasemide (Britomar) - round, biconvex, white to off-white tablets debossed SN with one side. 1 tablet contains active substance - torasemide 5 or 10 mg and excipients - guar gum, maize starch, anhydrous colloidal silica, magnesium stearate, lactose.
  Dosage scheme: per os, once a day, regardless of meals. The common starting dose in CHF - 10-20 mg once a day. If adequate diuretic effect is absent, the dose is increased approximately twofold up to adequate diuretic effect.
  Interventions: Drug: Prolonged release Torasemide (Britomar)
- Torasemide (Diuver) (Active Comparator): Torasemide (Diuver) - white to off-white, round, biconvex tablets. 1 tablet contain active substance - torasemide 5 or 10 mg and excipients - lactose monohydrate, maize starch, sodium glycolate starch, anhydrous colloidal silica, magnesium stearate. Dosage scheme: per os, once a day, after meals. Therapeutic dose - 5 mg a day. If necessary, a dose may be increased up to 20 mg a day, in some cases - up to 40 mg.
  Interventions: Drug: Torasemide (Diuver)

INTERVENTIONS:
Drug: Prolonged release Torasemide (Britomar)
  Arms: Prolonged release Torasemide (Britomar)
Drug: Torasemide (Diuver)
  Arms: Torasemide (Diuver)

SUMMARY:
Study hypothesis is that the time from randomization to the increase of natriuresis (%), time to standardization of natriuresis daily profile, blood pressure profile and the percentage reduction of central hemodynamic parameters will be relatively changed over the study period by more than 15%.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women in the age from 40 to 70 years.
2. Established diagnosis of II-III grade essential arterial hypertension
3. NYHA II-III chronic heart failure
4. Salt-sensitivity
5. Stable therapy for 3 months prior enrollment to the study including any diuretic, ACE-inhibitor, beta-blocker.
6. Signed informed consent for participation in the study.
7. Women with child-bearing potential should agree to use effective birth control methods from screening up to completion of the study, excluding situations when their sexual partner(s) are surgically sterilized, or whеn women do not have any sexual contacts. Effective methods of birth control are contraception methods which are used constantly and regularly (including implantable contraceptives, injectable contraceptives, oral contraceptives, transdermal contraceptives, intrauterine devices, diaphragms with spermicides, male or female condoms or cervical cap).

Exclusion Criteria:

1. Unlikely cooperation with a patient in the study period, disability
2. Identification of salt - resistance at screening
3. Patients that have had myocardial infarction, unstable angina pectoris, percutaneous coronary intervention heart failure, hypertensive encephalopathy, cerebrovascular accident (stroke) or transient ischaemic attack for the last 3 months.
4. Patients with severe heart failure (Stage IV of New York Heart Association), clinically significant aortic valve or mitral stenosis, uncorrected coarctation of the aorta, obstruction of cardiac output (obstructive hypertrophic cardiomyopathy)
5. Previous glomerulonephritis, severe pyelonephritis or another known severe renal disease which is confirmed by GFR < 40 ml/min/1.73 m2 calculated by Cockroft-Gault formula.
6. Secondary arterial hypertension, severe or uncontrolled AH at the study enrollment (BP> 180 mm Hg or DAP > 110 mm Hg)
7. Any severe, decompensated or unstable diseases or conditions which, on the investigator's opinion, endanger patient's life or aggravate disease prognosis (decompensated heart failure, anemia, severe diabetes mellitus, autoimmune, oncological diseases, hepatic, allergic reactions, connective tissue diseases, etc.)
8. Acute infectious diseases.
9. Hypersensitivity to components of Britomar or Diuver
10. Pregnancy, lactation period.
11. Participation in another clinical study for the last 30 days.
12. Scheduled coronary artery surgery (for example, stent implantation or coronary artery bypass grafting) or any other non-cardiological major surgery.
13. 13. Administration of drugs which affect natriuresis level (any diuretics which are not related with the study product). Patients are excluded from the study if they have taken the drugs for the last 48 years up to Visit D -10, in the screening period and/or treatment period/follow-up period of the study.
14. Use of narcotic drugs or alcohol abuse for the last 6 months and inability/unwillingness to refrain from narcotic drugs and excessive alcohol intake in the study period. The excessive alcohol intake is average alcohol >2 units of alcohol. A unit of alcohol for various beverages is 12 ounce (350 ml) of beer, 5 ounce (150 ml) of wine or 1.5 ounce (45 ml) of 80% alcohol.
15. Any other reason which would hinder patients' compliance with study requirements or their understanding of the study aim and potential risks of participation in study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Inflammatory markers excretion | 3 months
  15% or more increasing of the following Tamm-Horsfall protein, beta-2-microglobulin, osteoponin, TGF- β1 excretion in comperison with baseline level

SECONDARY OUTCOMES:
Daily sodium excretion | 3 months
  Increasing of daily sodium excretion on 30% or more in comparison with baseline
Augmentation index | 3 months
  Decreasing of augmentation index on 30 or more percents in comparison with baseline level
Albuminuria | 3 months
  Appearance of albuminuria of any stage or increasing of albuminuria level in case of existing albuminuria at the baseline. (measured by dipstick)

CONTACTS AND LOCATIONS:
Overall Officials: Grigory P Arutyunov, Prof, Principal Investigator — Russian Society for Heart Failure